CLINICAL TRIAL: NCT03610971
Title: Treatment Free Remission After Combination Therapy With Ruxolitinib Plus Tyrosine Kinase Inhibitors in Chronic Phase Chronic Myeloid Leukemia (CP-CML) Patients Who Relapsed After a Prior Attempt at TKI Discontinuation
Brief Title: Treatment Free Remission After Combination Therapy With Ruxolitinib Plus Tyrosine Kinase Inhibitors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: H. Jean Khoury Cure CML Consortium (Other); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19660; HJKC3-0002 (Other: H. Jean Khoury Cure CML Consortium)
Record Dates: First submitted 2018-07-19; First posted 2018-08-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia; Chronic Myeloid Leukemia, Chronic Phase
Keywords: CP-CML; Chronic Myeloid Leukemia; CML; combination therapy; BCR-ABL oncogene
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy + Remission Phase (Experimental): Combination therapy followed by treatment free remission (TFR) phase.
  Combination Therapy: Ruxolitinib plus BCR-ABL Tyrosine Kinase Inhibitors (TKIs).
  All eligible patients will begin ruxolitinib in combination with their BCR-ABL TKI on cycle 1 day 1 of the combination phase. For cycle 2 and beyond, if day 1 of a cycle is delayed, day 1 procedures should be repeated if out of the specified window and day 1 of the cycle is considered the day study drug is restarted. They will continue combination therapy for a total of 12 cycles. Each cycle will be approximately 28 days.
  At the end of 12 cycles ruxolitinib will be discontinued and any patient who has met the criteria for the treatment free remission (TFR) screening phase will enter into the TFR phase. Once in the TFR phase, participants will discontinue their BCR-ABL TKI and be monitored off treatment.
  Interventions: Drug: Ruxolitinib; Drug: BCR-ABL Tyrosine Kinase Inhibitor (TKI)

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib: 15 mg by mouth (PO) twice a day (BID).
  Other Names: Jakafi®
Drug: BCR-ABL Tyrosine Kinase Inhibitor (TKI) — The BCR-ABL TKIs that will be used include imatinib, dasatinib, nilotinib or bosutinib.
  Other Names: TKI

SUMMARY:
The purpose of this study is to determine if adding Ruxolitinib to a Tyrone Kinase Inhibitor (TKI), prior to a second attempt at stopping a TKI will lead to prolonged treatment free remission (TFR).

DETAILED DESCRIPTION:
All participants will have a confirmed diagnosis of chronic phase chronic myeloid leukemia (CML) and must have previously attempted to discontinue TKI therapy. All participants must be restarted on a TKI at the time of relapse in order to be eligible for this trial.

After completion of 12 cycles of combination therapy, eligible participants will remain in the TFR phase of the study for up to 36 months, and will have central polymerase chain reaction (PCR) testing during the first 24 months. Therefore, the total duration of the trial will be approximately 48 months (12 months on combination treatment phase + 36 months in the TFR phase).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Diagnosed with CML in chronic phase and have either the b3a2 (e14a2) or b2a2 (e13a2) variants that give rise to the p210 BCR-ABL protein.
* Must have a documented history of attempting only one prior TKI discontinuation under the guidance of a treating physician
* Must have met ALL the following criteria prior to first attempt to discontinue their TKI:

  * Stable molecular response (MR4; <0.01% IS) for > 2 years (allowance for a 2 week variance), as documented on at least 4 tests, performed at least 3 months apart. If any results are >0.05% IS, tests must have been repeated within 1 month and be less than 0.01% IS and stable.
  * Treatment with one of the following FDA approved TKI; imatinib, dasatinib, nilotinib or bosutinib, at any dose for a minimum of approximately 3 years (allowance of a 4 week variance) prior to discontinuing TKIs
  * Has been on any number of TKIs, but has not been resistant to any TKI (changes made for intolerance are allowed)
* Must have relapsed (defined as loss of major molecular response (MMR), RQ-PCR for BCR-ABL > 0.1% IS after first attempted discontinuation of TKI
* After first failed TFR attempt, must have a minimum duration of 1 year on a TKI, and must plan to remain on this same TKI for a minimum of 12 months during the combination treatment phase
* Current TKI must be the same as the TKI being taken prior to the initial TFR attempt (e.g., if patient is on imatinib prior to first TFR attempt, they should be on imatinib at time of enrollment on this study)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Must have a RQ-PCR for BCR-ABL less than 0.0032% IS (MR4.5) reported by the trial designated central lab at time of study enrollment
* Must adhere to all study contraception guidelines

Exclusion Criteria:

* History of accelerated or blast phase CML
* History of TKI resistance
* A second malignancy requiring active treatment
* Have previously received treatment with a JAK inhibitor.
* Platelet count less than 100 × 10^9/L or an absolute neutrophil count of less than 1 × 10^9/L or Hemoglobin less than 8 g/dL
* AST and ALT ≥ 3 times the institutional upper limit of normal (ULN)
* Creatinine ≥ 2 times ULN
* Total bilirubin ≥ 1.5 times ULN or >3.0 x the ULN with Gilbert Syndrome (unless direct bilirubin is within normal limits)
* Pregnant or lactating
* Unable to comply with lab appointments schedule and patient response outcome assessments
* Another investigational drug within 4 weeks of enrollment
* Any serious medical or psychiatric illness that could, in the investigator's opinion, interfere with the completion of treatment according to this protocol
* Have undergone a prior allogeneic transplant
* Screening 12-lead ECG showing a baseline corrected QT interval >500msec (patients with a pacemaker will still be eligible with QTc>500msec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
12 Month Treatment Free Remission (TFR) | 12 months post 12 cycles of treatment
  TFR rate after completion of 12 cycles of combination therapy.

SECONDARY OUTCOMES:
Adverse Events Possibly Related to Study Treatment | Up to 30 days post treatment, approximately 13 months per participant
  Establish the adverse event profile of ruxolitinib in combination with BCR-ABL TKIs: Adverse Events (AEs) and Serious Adverse Events (SAEs) according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0, that are possibly, probably, or definitely related to study treatment.

OTHER OUTCOMES:
Incidence of Improved Scores in Health Related Quality of Life Questionnaire | Up to 48 months
  Number of participants with an improved score in 2 or more categories of the questionnaire at the end of the TFR phase, when compared to the score for the same questions when completed at the end of 12 cycles of combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pinilla-Ibarz, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory -Winship Cancer Institute, Atlanta, Georgia
  - Memorial Sloan Kettering - Bergen, Montvale, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin